CLINICAL TRIAL: NCT06468891
Title: Analyzing Gait Parameters Among Women With and Without Stress Urinary Incontinence
Acronym: GPWSUI
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, Cairo University, Cairo University
Other Study IDs: KFSIRB200- 249
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Gait; Stress Urinary Incontinence; Women
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with stress urinary incontinence: This group includes 62 participants with chronic stress urinary incontinence.
  Interventions: Other: Incontinence Symptom Severity Index; Other: Force platform; Other: The STT three-dimensional motion analysis (3DMA) system
- women without stress urinary incontinence: This group includes 62 participants who are free from urinary incontinence symptoms and pelvic floor dysfunction.
  Interventions: Other: Incontinence Symptom Severity Index; Other: Force platform; Other: The STT three-dimensional motion analysis (3DMA) system

INTERVENTIONS:
Other: Incontinence Symptom Severity Index — * The ISSI consists of eight items that assess different aspects of urinary incontinence symptoms, including emptying difficulties, nocturia, daytime frequency, stress incontinence, urge incontinence, leakage with activity, and pad use.
  * Each item is scored on a scale of (0 to 3) or (0 to 4), depending on the severity of the symptom. Higher scores indicate more severe symptoms.
  * The total ISSI score is obtained by summing the scores of all eight items, resulting in a range of 0 to 32 or 0 to 40, depending on the version used.
  * The severity of urinary incontinence symptoms can be categorized based on the total ISSI score
  Other Names: (ISSI).
Other: Force platform — Use the provided software or tools to analyze the recorded force data, including Step Cycle Duration (ms), Time of Contact (ms), Swing Duration (ms), Single Step Duration (ms), Double Support Duration (ms), Initial Contact (ms) , Loading Response (ms), Mid Stance (ms), Terminal Stance (ms), Step Cycle Length, Half Step Length for left and right lower limbs.
  * Interpret the data to draw conclusions about the forces exerted during the subject's movements or activities.
Other: The STT three-dimensional motion analysis (3DMA) system — The STT three-dimensional motion analysis (3DMA) system (STT Systems Company, Zuatzu Business Park, Easo Building, 2nd Floor, San Sebastián, Spain) was used for the assessment of spatiotemporal characteristics of gait. It is an indoor optical system that consists of four cameras, fifteen markers, and computer software for automatic three-dimensional motion capture and analysis. CLINICAL 3DMA V.6.11 is professional software with highly accurate marker tracking. The STT Helen Hayes protocol was used for the gait analysis in this study.

SUMMARY:
This study will contribute to the existing body of knowledge on stress urinary incontinence and its impact on gait. The findings may have implications for the development of targeted interventions and rehabilitation strategies to improve mobility and quality of life in women with stress urinary incontinence

DETAILED DESCRIPTION:
Use the provided software or tools to analyze the recorded data, including (cadence, velocity, swing, and double limb support, stride time, step length, and stride length) of gait. The software measures the cadence as total number of steps per minute, and it measures the stride time as the time (in sec) from heel strike of one limb to the next heel strike of the same limb. Also, the software measures the duration of stance, swing, and double limb support as percentage of stride time. Also, the software measures the step and stride length (in cm).

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-60 years old.
* Women with BMI ≥30.
* Women are free from any other gynecological disorders or symptoms that may affect the results of the study.
* All participants who will be enrolled in the study sign the informed consent form.
* All participants will be of multiparas.
* All participants will be diagnosed with a mild degree of stress urinary incontinence.

Exclusion Criteria:

* Pregnancy
* Neurological Disorders: such as Parkinson's disease , multiple sclerosis, or any neurological dysfunction that may affect the gait parameters
* Musculoskeletal disorders: such as severe osteoarthritis or lower limb amputations
* Significant cognitive impairment: or dementia
* Previous pelvic surgery as pelvic organ prolapse repair or anti-incontinence procedures.
* Other significant medical conditions that could affect gait include severe cardiovascular disease or severe respiratory conditions.
* Walking pain.

Ages: 40 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: One hundred twenty-four female participants who have stress urinary incontinence will participate in this study. Their ages will be ranged from 40 to 60 years. The participants will be selected from Mansoura University Hospitals and randomly distributed into two equal groups in numbers.
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Incontinence Symptom Severity Index | one day
  The Incontinence Symptom Severity Index (ISSI) is a self-assessment instrument used to measure the severity of female urinary storage and voiding symptoms.

SECONDARY OUTCOMES:
Force platform | one day
  After data collection, the recorded data is analysed to extract various gait parameters. These parameters include: Srtide lengh for left and right lower limbs, Srtide time for left and right lower limbs, Step Cycle Duration (ms), Time of Contact (ms), Swing Duration (ms), Double Support Duration (ms).The findings from the gait analysis are typically documented in a report to be used for statistical analysis.
The STT three-dimensional motion analysis (3DMA) system | one day
  The STT three-dimensional motion analysis (3DMA) system (STT Systems Company, Zuatzu Business Park, Easo Building, 2nd Floor, San Sebastián, Spain) was used for the assessment of spatiotemporal characteristics of gait. It is an indoor optical system that consists of four cameras, fifteen markers, and computer software for automatic three-dimensional motion capture and analysis. CLINICAL 3DMA V.6.11 is professional software with highly accurate marker tracking. The STT Helen Hayes protocol was used for the gait analysis in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elabd OM, Etoom M, Jahan AM, Elabd AM, Khedr AM, Elgohary HM. The Efficacy of Muscle Energy and Mulligan Mobilization Techniques for the Upper Extremities and Posture after Breast Cancer Surgery with Axillary Dissection: A Randomized Controlled Trial. J Clin Med. 2024 Feb 8;13(4):980. doi: 10.3390/jcm13040980. PMID 38398293
- See also: research paper — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10889574/